CLINICAL TRIAL: NCT03882073
Title: A Novel Approach to Upper Extremity Amputation to Augment Volitional Control and Restore Proprioception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Carty, Director, Lower Extremity Transplant Program, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018p001893; CDMRP-170384 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Modified amputation procedure
  Interventions: Procedure: Modified amputation procedure
- Control group (Active Comparator): Standard amputation procedure
  Interventions: Procedure: Standard amputation procedure

INTERVENTIONS:
Procedure: Modified amputation procedure — A fishmouth incision will be made. Radial and ulnar (BEA) or humoral (AEA) osteotomies will be performed. Segments of the flexor carpi radialis (FCR), extensor carpi radialis longus (ECRL), flexor digitorum profundi (FDP), extensor digitorum communis (EDC), flexor pollicis longus (FPL) and extensor pollicis longus (EPL) will be isolated, as well as the biceps (B) and triceps (T) groups in the AEA model; if it is not possible to preserve native innervation to these muscles, functional motor units will be constructed from muscle coapted to the appropriate motor nerve endings. Sensory nerve endings of the distal median, ulnar and radial nerves will then be isolated and redirected to discrete skin patches in the proximal residual forearm or proximal brachium. Coaptation of the FCR/ECRL, FDP/EDC, FPL/EPL and B/T muscles will then be performed to promote dynamic coupling of these agonist/antagonist pairs. The skin envelope will then be closed in layers over percutaneous drains.
  Arms: Intervention group
Procedure: Standard amputation procedure — Amputation is performed via standard techniques at either the BEA or AEA level. No construction of agonist-antagonist muscle pairs will be performed.
  Arms: Control group

SUMMARY:
The hypothesis of this research protocol is that the investigators will be able to redesign the manner in which upper limb amputations are performed so as to enable volitional control of next generation prosthetic devices and restore sensation and proprioception to the amputated limb. The investigators will test this hypothesis by performing modified above elbow or below elbow amputations in ten intervention patients, and compare their outcomes to ten control patients who have undergone tradition amputations at similar levels. The specific aims of the project are:

1. To define a standardized approach to the performance of a novel operative procedure for both below elbow (BEA) and above elbow amputations (AEA)
2. To measure the degree of volitional motor activation and excursion achievable in the residual limb constructs, and to determine the optimal configuration and design of such constructs
3. To describe the extent of proprioceptive feedback achievable through the employment of these modified surgical techniques
4. To validate the functional and somatosensory superiority of the proposed amputation technique over standard approaches to BEA and AEA
5. To develop a modified acute postoperative rehabilitation strategy suited to this new surgical approach

This will be a phase I/pilot clinical trial to be performed over a three-year period as a collaborative initiative involving Brigham & Women's Hospital/Brigham & Women's Faulkner Hospital (BWH/BWFH), Walter Reed National Military Medical Center (WRNMMC), and the Massachusetts Institute of Technology (MIT). The investigators will plan to perform 6 of the 10 amputations at BWH/BWFH, and 4 of the amputations at WRNMMC.

DETAILED DESCRIPTION:
Upper extremity amputation is among the oldest known surgical procedures in medical history, with many of its technical principles having first been elucidated by Hippocrates. Despite the passage of more than two millennia, relatively little has changed in the operative approach to upper limb sacrifice. An estimated 58,000 patients in the United States currently suffer from upper extremity limb loss at either the above elbow (AEA) or below elbow (BEA) level, and the prevalence of upper limb amputation is expected to rise to approximately 95,000 patients by 2050.

Normal function of the upper limb is enabled through the dynamic interplay of multiple muscle groups acting in concert. Manual dexterity is a remarkably orchestrated biomechanical process that is dependent upon a complex feedback loop involving the central and peripheral nervous systems and the musculoskeletal system. In their native state, the muscles of the upper extremity exist in a balanced agonist/antagonist situation in which volitional activation of one muscle leads not only to its contracture, but also to passive stretch of its opposite. Changes in muscle tension manifest through this interaction of agonist and antagonist units lead to stimulation of specialized receptors within the muscle fibers (e.g., muscle spindle fibers and Golgi tendon organs) that transmit joint position information to the cerebral cortex. Such feedback, in conjunction with cutaneous sensory information from skin mechanoreceptors, provides us with a sense of limb proprioception that ultimately enables high fidelity limb control, even in the absence of visual feedback.

Unfortunately, the standard operative approach to upper limb amputation at either the AEA or BEA level obliterates many of the dynamic relationships characteristic of the uninjured upper extremity. Initial surgical exposure is typically accomplished through a fishmouth-pattern incision, followed by progressive transection of muscles, vessels, nerves and bone at the level of the incision. Tissues distal to the site of structural transection are discarded, regardless of whether or not there may be viable segments, and the proximal residual muscles are layered over the distal transected bone in order to provide insulation to this exposed osseous surface. The surrounding skin is then advanced over the bone/muscle construct in order to achieve definitive closure. The rudimentary approximation of discordant tissues in the distal limb in this approach results in a disorganized scar mass in which normal dynamic muscle relationships are destroyed. The uncoupling of native agonist/antagonist muscle pairings results in isometric contraction of residual muscle groups upon volitional activation, producing incomplete, unbalanced neural feedback to the brain that results in aberrant perception of residual limb position. Such disturbed feedback not only leads to impaired limb function with prostheses, but also manifests as pathological sensory perception of the extremity in the form of phantom limb and phantom pain symptoms.

To date, the limitations of these approaches have been tolerated due to the fairly simplistic goal of upper limb amputation: to provide a stable, padded surface for mounting a prosthesis. Historically, upper limb prostheses have afforded amputees the opportunity to recover at least some measure of upper limb function. However, such devices have generally not been able to recapitulate the complex biomechanics of the human upper limb due to limited ranges of motion and lack of feedback control. These limitations have resulted in reported upper limb prosthesis rejection rates ranging from 23% to 45%, including both body-powered and myoelectric devices.

However, the capabilities of modern prostheses are now expanding remarkably. Technological advances including increasingly miniaturized electronics, wireless communications and ever-refined positional sensors have enabled prosthetic developers to create next-generation bionic limbs with greatly enhanced degrees of freedom over prior models. Even more advanced prostheses are currently being developed that have the potential to offer sensory feedback - both tactile and positional - in a manner never before seen. Such prosthetic devices, while not yet available commercially, are presently being studied in experimental settings. For example, the Defense Advanced Research Projects Agency (DARPA) recently issued a request for proposals under the Hand, Proprioception and Touch Interfaces (HAPTIX) Program incorporating an upper limb prosthesis including six degrees of freedom at the wrist, thumb and all digits, 10 pressure sensors capable of providing sensory feedback, and joint angle and velocity sensors capable of providing joint position data.

Despite these technological advances in prosthesis development, surgical methods regarding management of the residual limb have not kept pace with these enhanced prosthesis capabilities. Classic techniques of upper limb amputation do not provide innervated interfaces that can serve as relays for complex prosthetic control; without such biological actuators in the residual limb to provide afferent and efferent conduits for information exchange, next generation prostheses are of little use. Stated another way, next generation prosthetic devices currently incorporate drivers and sensors capable of providing far more enhanced functionality than ever before seen, but standard approaches to limb amputation do not deliver a way to effectively link these prosthetics to their intended beneficiaries. An evolution in the manner in which upper limb amputations are performed - one that will provide a biological interface that will allow upper limb amputees to take advantage of the enhanced capabilities offered by the remarkable prostheses currently under development - is now required.

Recognition of the increased need for effective neural interfaces for prosthetic limbs can be seen in the expanding number of efforts in this sphere over the past decade. Initial efforts to provide high-resolution control of distal prostheses were focused primarily on indirect and direct brain interfaces, either through placement of electroencephalographic scalp sensors or implantable parenchymal electrodes, respectively. However, such endeavors have been plagued by poor resolution, inconsistencies in signal acquisition and, in the case of implantable devices, progressive foreign body reactions leading to impulse degradation over time.

As the limitations of brain interfaces have become more evident, focus has shifted instead to peripheral control loci. Efforts in this vein have included direct peripheral nerve interfaces including interposed sieves and cuffs designed to transduce electrical signals directly from individual nerve fascicles to distal prostheses. Such monitors have, however, shown little clinical promise due to progressive nerve compression secondary to scarring, as well as to significant neurological crosstalk and interference in biological models.

The most promising efforts regarding peripheral nerve interface development are now within the realm of biological systems. These models consist of configurations in which native tissues are innervated with distal nerve endings to create biological actuators for distal prosthesis control and feedback. The two leading models in this sphere are as follows:

* Targeted Muscle Re-innervation (TMR): Pioneered by Dumanian and Kuiken et al, TMR is a technique whereby a series of nerve transfers is used to re-innervate specific target muscles to create additional prosthesis control sites after distal limb amputation.
* Regenerative Peripheral Nerve Interfaces (RPNI): Championed by Cederna et al, RPNI offers an alternative version of an innervated biological interface. An RPNI is a surgical construct that consists of a non-vascularized segment of muscle that is coapted to a distal motor or sensory nerve ending.

While both TMR and RPNIs have demonstrated promise in offering improved functionality to patients who have already undergone amputation, neither technique has been incorporated into a fundamental redesign of the way in which amputations are performed in the first place; in all cases of clinical implementation of TMR or RPNIs reported to date in the literature, these techniques have been employed to further optimize the functionality of patients who had already experienced limb loss.

The clinical protocol proposes a reinvention of the manner in which upper limb amputations are performed, building upon several of the principles established in the work already performed in the realm of TMR and RPNIs. As elaborated below, the core innovation is the utilization of distal limb tissues that would ordinarily be sacrificed in the course of standard lower limb amputations to provide the substrate for natively innervated pairings of agonist/antagonist muscles capable not only of intuitive, volitional motor activation but also proprioceptive feedback. Conceptually, this idea consists of physical linkage of biologically opposed muscles (e.g., the biceps and triceps) such that when neurologically triggered contraction of one muscle is effected, simultaneous stretch of its partner is also achieved, resulting in observable motion of the dyad and stimulation of standard proprioceptive pathways. The investigators have named this construct the agonist-antagonist myoneural interface (AMI).

The manner in which this dynamic agonist/antagonist muscle concept may be operationalized clinically depends upon whether or not intact, innervated and vascularized native muscles are present at the time of operative intervention. Over the past five years, the research group has developed experimental models for a variety of clinical scenarios through a series of preclinical investigations in both murine and caprine populations.

If healthy native muscle is available as a reconstructive substrate, coaptation of the distal ends of disinserted agonist/antagonist pairs may be incorporated into the design of the residual limb; when coupled with a native synovial canal as a gliding interface, a pulley-like system can be established to provide a dynamic muscle construct. Construction of AMIs in a rat model have demonstrated preservation of construct muscle bulk, viability over time and production of graded afferent signals in response to ramp and hold stretches in a manner similar to native muscle architecture. Furthermore, performance of an amputation at the transtibial level with incorporation of AMI construction in a goat model has demonstrated clear coupled motion of the agonist-antagonist pair in the presence of both natural neural commands and artificial muscle stimulation.

Based on these proof of concept animal studies, the investigators hypothesize that the AMI offers the potential to provide a biological relay for volitional control that is superior to other neural interface strategies, with the additional benefit of being able to restore limb proprioception. When coupled with an appropriately adapted next-generation prosthesis, the AMI thus may provide the first biological mechanism to achieve true closed-loop neural interactivity with a mechanical limb.

The investigators here propose a three-year, prospective, controlled assessment of the functional and somatosensory advantages of the modified amputation model in an upper extremity scenario. The investigators believe this model has the potential to provide upper limb amputees with a biological interface that offers not only unprecedented, high-resolution motor control of prostheses, but also is highly intuitive and capable of restoring limb proprioception. If manifest, these augmented capabilities may result in improved functionality and overall health outcomes, including more robust return to work status and diminished psychological strain.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 65
* Candidates for elective unilateral or bilateral upper extremity amputation at either the above elbow or below elbow level due to traumatic injury, congenital limb deformities or progressive arthritis
* Must demonstrate sufficiently sound health to undergo the operative procedure, including adequate cardiopulmonary stability to undergo general anesthesia (specifically, American Society of Anesthesiology Class I or II)
* Must have intact inherent wound healing capacity
* Must demonstrate adequate communication skills to convey the status of their sensorimotor recovery throughout the postoperative phase,
* Must exhibit proper level of motivation to comply with postoperative follow up requirements
* Must be willing to also consent to study activities taking place at Massachusetts Institute of Technology (approved under same IRB protocol via ceded IRB review) as some outcome measures will be assessed at that site

Exclusion Criteria:

* Patients beyond the stated age restrictions
* Those with severe illness rendering them unable to undergo the operative procedure safely (e.g., unresolved sepsis or cardiopulmonary instability manifest as documented coronary artery disease and/or chronic obstructive pulmonary disease)
* Patients with active infections, particularly deep infections in the arm to be amputated
* Patients who are taking immunosuppressive agents
* Patients with impairment in inherent wound healing pathways, such as those with primary connective tissue disorders or those on chronic steroid therapy
* Patients with extensive peripheral neuropathies (diabetic or otherwise) that would potentially inhibit appropriate reinnervation of the surgical constructs
* Active smokers; those patients willing to undergo tobacco cessation will need to be completely abstinent from tobacco use for at least 6 weeks preoperatively
* Patients who are unable to provide informed consent and those with a demonstrated history of poor compliance
* Pregnant women will not be considered due to the potential risks of general anesthesia

Patients will not be excluded from participation in the study on the grounds of minority status, religious status, race or gender. Non-English speaking patients will not be excluded from the study; interpreters will be made available to them for translation of both verbal interactions and written documents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Motor Unit Innervation | 0-36 months
  Intact volitional activation of motor constructs, as assessed by electromyographic evidence of activation (muscle potentials measured in mV)
Motor Unit Excursion | 0-36 months
  Intact volitional activation of motor constructs with measurable excursion, as assessed by ultrasound (excursion measured in mm)
Proprioception Recovery | 0-36 months
  Manifestation of functional proprioception with motor unit activation, as evidenced by spatial limb position testing using a modified upper limb prosthesis (accurate limb positioning relative to target measured in mm)

SECONDARY OUTCOMES:
Infection Rate | 0-36 months
  Postoperative infection rate
Delayed Wound Healing Rate | 0-36 months
  Postoperative delayed wound healing rate
Operative Revision Rate | 0-36 months
  Subsequent rate of reoperation
Seroma Rate | 0-36 months
  Postoperative seroma rate
Deep Vein Thrombosis Rate | 0-36 months
  Postoperative deep vein thrombosis rate
30-Day Mortality Rate | 0-36 months
  Postoperative 30-day mortality rate
General Health Status | 0-36 Months
  Preoperative and postoperative general health status, as assessed by four validated surveys
Muscle Atrophy | 0-36 Months
  Postoperative muscle atrophy, as evidenced by changes in muscle volume
Sensory Recovery | 0-36 Months
  Postoperative sensory recovery, as assessed by cutaneous stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carty, MD, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology Media Lab, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No
No plan for individual participant data sharing

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Biddiss EA, Chau TT. Upper limb prosthesis use and abandonment: a survey of the last 25 years. Prosthet Orthot Int. 2007 Sep;31(3):236-57. doi: 10.1080/03093640600994581. PMID 17979010
- [Background] Schultz AE, Kuiken TA. Neural interfaces for control of upper limb prostheses: the state of the art and future possibilities. PM R. 2011 Jan;3(1):55-67. doi: 10.1016/j.pmrj.2010.06.016. PMID 21257135
- [Background] Shih JJ, Krusienski DJ, Wolpaw JR. Brain-computer interfaces in medicine. Mayo Clin Proc. 2012 Mar;87(3):268-79. doi: 10.1016/j.mayocp.2011.12.008. Epub 2012 Feb 10. PMID 22325364
- [Background] Kung TA, Bueno RA, Alkhalefah GK, Langhals NB, Urbanchek MG, Cederna PS. Innovations in prosthetic interfaces for the upper extremity. Plast Reconstr Surg. 2013 Dec;132(6):1515-1523. doi: 10.1097/PRS.0b013e3182a97e5f. PMID 24281580
- [Background] Navarro X, Krueger TB, Lago N, Micera S, Stieglitz T, Dario P. A critical review of interfaces with the peripheral nervous system for the control of neuroprostheses and hybrid bionic systems. J Peripher Nerv Syst. 2005 Sep;10(3):229-58. doi: 10.1111/j.1085-9489.2005.10303.x. PMID 16221284
- [Background] Dumanian GA, Ko JH, O'Shaughnessy KD, Kim PS, Wilson CJ, Kuiken TA. Targeted reinnervation for transhumeral amputees: current surgical technique and update on results. Plast Reconstr Surg. 2009 Sep;124(3):863-869. doi: 10.1097/PRS.0b013e3181b038c9. PMID 19730305
- [Background] Kuiken TA, Li G, Lock BA, Lipschutz RD, Miller LA, Stubblefield KA, Englehart KB. Targeted muscle reinnervation for real-time myoelectric control of multifunction artificial arms. JAMA. 2009 Feb 11;301(6):619-28. doi: 10.1001/jama.2009.116. PMID 19211469
- [Background] Clites TR, Carty MJ, Srinivasan S, Zorzos AN, Herr HM. A murine model of a novel surgical architecture for proprioceptive muscle feedback and its potential application to control of advanced limb prostheses. J Neural Eng. 2017 Jun;14(3):036002. doi: 10.1088/1741-2552/aa614b. Epub 2017 Feb 17. PMID 28211795
- [Background] Clites TR, Carty MJ, Ullauri JB, Carney ME, Mooney LM, Duval JF, Srinivasan SS, Herr HM. Proprioception from a neurally controlled lower-extremity prosthesis. Sci Transl Med. 2018 May 30;10(443):eaap8373. doi: 10.1126/scitranslmed.aap8373. PMID 29848665
- [Background] Taghipour H, Moharamzad Y, Mafi AR, Amini A, Naghizadeh MM, Soroush MR, Namavari A. Quality of life among veterans with war-related unilateral lower extremity amputation: a long-term survey in a prosthesis center in Iran. J Orthop Trauma. 2009 Aug;23(7):525-30. doi: 10.1097/BOT.0b013e3181a10241. PMID 19633463
- [Background] Lipsitz SR, Fitzmaurice GM, Orav EJ, Laird NM. Performance of generalized estimating equations in practical situations. Biometrics. 1994 Mar;50(1):270-8. PMID 8086610